CLINICAL TRIAL: NCT06097416
Title: A Phase III, Multi-institutional Randomised Trial Comparing Neoadjuvant Chemoradiotherapy (NARCT) and Total Neoadjuvant Therapy (TNT) in Patients With T3 (a/b/c) Rectal Cancer
Brief Title: Neoadjuvant Chemoradiotherapy Versus Total Neoadjuvant Therapy in the Treatment of T3 Rectal Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: St. James's Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Michael Kelly, Consultant Colorectal Surgeon, St. James's Hospital, Ireland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: St. James's Hospital
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Neoadjuvant chemoradiotherapy; Total neoadjuvant therapy; Survival
MeSH Terms: conditions — Rectal Neoplasms | interventions — Neoadjuvant Therapy; Trinitrotoluene

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neoadjuvant chemoradiotherapy (Active Comparator): The NARCT regimen is prescribed specifically as standard 5-FU over several weeks. The CRT regimen consists of the standard algorithms: a total of 5400-5600 cGy of radiation (4500 cGy to the pelvis, with an integrated boost to the primary tumour and involved nodes of 500 cGy followed by an option boost to the primary tumour and involved nodes) delivered in 27-28 fractions, respectively, of 180-200 cGy each over a 5-6 week period.
  Interventions: Drug: Neoadjuvant Chemoradiotherapy
- Total Neoadjuvant Therapy (Active Comparator): Sequence of TNT regimen can be classified as induction (chemotherapy first) or consolidation (radiation first) treatment. All patients received the same chemotherapy (FOLFOX) and long-course chemoradiotherapy (50.4 Gy in 28 fractions) before surgery. However timing of TNT can differ depending on concerns of local and distal failure.
  Interventions: Drug: Total Neoadjuvant Therapy

INTERVENTIONS:
Drug: Neoadjuvant Chemoradiotherapy — 5-FU is a fluoropyrimidine antimetabolite considered to act primarily as an inhibitor of thymidylate synthase. 5-FU is supplied as a colourless-to-faint yellow solution in 10-mL single use vials. Each 10 mL of solution contains 500 mg 5-FU, with pH adjusted to approximately 9.2 with sodium hydroxide.
  The CRT regimen consists of the standard algorithms: a total of 5400-5600 cGy of radiation (4500 cGy to the pelvis, with an integrated boost to the primary tumour and involved nodes of 500 cGy followed by an option boost to the primary tumour and involved nodes) delivered in 27-28 fractions, respectively, of 180-200 cGy each over a 5-6 week period.
  Other Names: NACRT
  Arms: Neoadjuvant chemoradiotherapy
Drug: Total Neoadjuvant Therapy — 5-FU is a fluoropyrimidine antimetabolite considered to act primarily as an inhibitor of thymidylate synthase. 5-FU is supplied as a colourless-to-faint yellow solution in 10-mL single use vials. Each 10 mL of solution contains 500 mg 5-FU, with pH adjusted to approximately 9.2 with sodium hydroxide.
  Oxaliplatin is an organoplatinum complex in which the platinum atom is complexed with 1,2- diaminocyclohexane with an oxalate ligand as a leaving group. Platinum content is 48.1% to 50.1%.
  All patients received the same chemotherapy (FOLFOX) and long-course chemoradiotherapy (50.4 Gy in 28 fractions) before surgery.
  Other Names: TNT
  Arms: Total Neoadjuvant Therapy

SUMMARY:
The gold standard treatment for locally advanced, non-metastatic rectal cancer includes neoadjuvant chemoradiotherapy (NACRT), total mesorectal excision (TME) and adjuvant chemotherapy (AC). The primary goal of treatment is to achieve local disease control, reduce tumour volume and minimise the risk of distant metastases. While this multimodal treatment approach has offered improvements in local control and sphincter preservation, it has had little effect on distant recurrence and overall survival. We aim to compare NACRT and TME using the following endpoints:

Primary -->To compare the effects neoadjuvant chemoradiotherapy versus total neoadjuvant therapy (TNT) for T3 rectal cancer on overall survival.

Secondary --> To compare the effects neoadjuvant chemoradiotherapy (NARCT) and total neoadjuvant therapy (TNT) for cT3 rectal cancer on clinical outcomes:

* Clinical complete response (cCR)
* Pathological complete response (pCR)
* Disease-free survival (DFS)
* Organ preservation
* Overall morbidity / mortality
* Treatment-related morbidity / mortality
* Peri-operative outcomes

ELIGIBILITY:
Patients are eligible to be included in the study only if they meet all of the following criteria:

1. Written informed consent must be given according to ICH/GCP and national/local regulations and be obtained prior to any study-related procedures.
2. Histologically or cytologically confirmed surgically resectable adenocarcinoma of the rectum.
3. Clinical stage II (T3, N-) \
4. Absence of metastatic disease
5. Eastern Co-operative Oncology Group (ECOG) performance status > 2.
6. Age > to 18.
7. Estimated life expectancy ≥ 12 months.
8. No active infections requiring systemic antibiotic treatment (oral antibiotics are acceptable at the discretion of the treating physician).
9. Measurable disease, as defined by RECIST Version 1.1
10. Adequate haematological, hepatic, and renal function defined as:

    a. Renal: i. Calculated creatinine clearance (CrCl) > 50ml/min (see Appendix G)

    b. Liver function tests: i. Total Bilirubin < 1.5 ULN

    (OR < 3 x ULN (< Grade 2) in the presence of documented Gilbert's syndrome (unconjugated hyperbilirubinemia) or liver metastases at baseline.) ii. ALT and AST < 2.5 x ULN (< 5 x ULN with liver involvement of their cancer) iii. Alkaline Phosphatase < 2.5 x ULN (< 5 x ULN with liver involvement of their cancer)

    c. Haematology: i. Haemoglobin > 9 g/dL (< Grade 1) ii. Absolute neutrophil count > 1.5 x 109/L iii. Platelet count > 100 x109/L (≤ Grade 1)
11. Normal thyroid function defined as a TSH within normal local institutional range
12. Able to swallow and retain oral medication
13. Women of childbearing potential (WOCBP) and male patients with partners of childbearing potential; agree to remain abstinent (refrain from heterosexual intercourse) or use highly effective contraception measures during the treatment period. For women, highly effective contraception should be used, for X months after last dose of (INSERT AGENT). For men, highly effective contraception should be used, for X months after (INSERT AGENT). (Highly effective contraception is defined in the study as methods that achieve a failure rate of less than 1% per year when used consistently and correctly. Such methods include:

    i. Combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal).

    ii. Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable and implantable).

    iii. Intrauterine device (IUD). iv. Intrauterine hormone-releasing system (IUS). v. Bilateral tubal occlusion. vi. Successfully vasectomised partner. vii. Sexual abstinence.)
14. Women of childbearing potential must have pregnancy excluded by urine or serum beta-HCG testing within 7 days prior to registration.

Exclusion criteria:

Patients who meet any of the following criteria at the time of screening will be excluded from study registration:

1. Received prior chemotherapy for local or metastatic disease.
2. Locally advanced rectal cancer; >T3, Nodal disease
3. Primary unresectable rectal cancer. A tumour is considered unresectable when invading adjacent organs and an en bloc resection will not achieve negative margins.
4. Received prior pelvic radiotherapy.
5. Patients unable to undergo MRI.
6. Previous or concurrent active malignancy ≤ 5 years prior to registration with the exception of non-melanotic skin cancer or carcinoma in situ of any type, or other cancers that the treating Investigator does not feel will impact the study objectives.
7. Screening electrocardiogram (ECG) with evidence of:

   1. QT prolongation (QTc > 450ms in males and > 470ms in females)
   2. Clinically significant cardiac arrhythmias, complete left bundle branch block, high atrioventricular AV block (e.g. bi-vascular block , Mobitz type II and third degree AV block
   3. Other severe cardiac dysfunction

   (ECG must be assessed for all patients within 14 days prior to registration).
8. Clinically significant cardiovascular disease including:

   1. Cerebrovascular accident within 6 months prior to registration
   2. Myocardial infarction within 6 months prior to registration
   3. Uncontrolled angina
   4. Uncontrolled or poorly controlled arterial hypertension (i.e. BP >150/90mmHg under treatment with at a maximum three antihypertensive drugs)
   5. Clinically significant valvular disease
   6. Congestive Heart Failure (NYHA > Class 2 (See Appendix E)
   7. Known family history of idiopathic cardiac arrest or sudden death whereby a cardiac cause cannot be excluded
   8. Known history or family history of Brugada Syndrome.
9. Known pulmonary compromise, as determined by the treating investigator, resulting from intercurrent pulmonary illness, but not limited to, any pulmonary disorder (e.g. severe asthma, severe chronic obstructive pulmonary disease (COPD), restrictive lung disease.
10. Creatinine level >1.5x ULN
11. Patients with a history of any arterial thromobotic event within the past 6 months. This includes angina (stable or unstable), MI, TIA or CVA.
12. Patients with a history of venous thrombotic episodes such as DVT, PE occurring more than 6 months prior to enrolment may be considered for protocol participation, provided they are on stable doses of anticoagulant therapy. Similarly, patients who are anticoagulated for atrial fibrillation or other conditions may participate, provided they are on stable doses of anticoagulant therapy.
13. Pregnant or nursing women.
14. Concurrent treatment with any other investigational agents within 30 days prior to registration.
15. Any psychological, physical, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; (those conditions should be discussed with the patient before registration in the trial).
16. Unable or unwilling to discontinue (and substitute if necessary) use of prohibited medications for at least 30 days prior to and for the duration of study treatment (see section 7.5 for a description of prohibited medications).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Five years
  Alive

SECONDARY OUTCOMES:
Clinical complete response | 6 months
  No residual tumour visible on imaging
Pathological complete response | 6 months
  Absence of residual invasive or in situ tumour on biopsy / resected specimen.
Disease-free survival | 5 years
  Measure of time after treatment where no evidence of disease is found.
Progression-free survival | 5 years
  Time from randomisation to occurrence of disease progression or death

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sauer R, Becker H, Hohenberger W, Rodel C, Wittekind C, Fietkau R, Martus P, Tschmelitsch J, Hager E, Hess CF, Karstens JH, Liersch T, Schmidberger H, Raab R; German Rectal Cancer Study Group. Preoperative versus postoperative chemoradiotherapy for rectal cancer. N Engl J Med. 2004 Oct 21;351(17):1731-40. doi: 10.1056/NEJMoa040694. PMID 15496622
- [Background] Kong JC, Soucisse M, Michael M, Tie J, Ngan SY, Leong T, McCormick J, Warrier SK, Heriot AG. Total Neoadjuvant Therapy in Locally Advanced Rectal Cancer: A Systematic Review and Metaanalysis of Oncological and Operative Outcomes. Ann Surg Oncol. 2021 Nov;28(12):7476-7486. doi: 10.1245/s10434-021-09837-8. Epub 2021 Apr 23. PMID 33891203
- [Background] Feeney G, Sehgal R, Sheehan M, Hogan A, Regan M, Joyce M, Kerin M. Neoadjuvant radiotherapy for rectal cancer management. World J Gastroenterol. 2019 Sep 7;25(33):4850-4869. doi: 10.3748/wjg.v25.i33.4850. PMID 31543678
- [Background] Hoendervangers S, Burbach JPM, Lacle MM, Koopman M, van Grevenstein WMU, Intven MPW, Verkooijen HM. Pathological Complete Response Following Different Neoadjuvant Treatment Strategies for Locally Advanced Rectal Cancer: A Systematic Review and Meta-analysis. Ann Surg Oncol. 2020 Oct;27(11):4319-4336. doi: 10.1245/s10434-020-08615-2. Epub 2020 Jun 10. PMID 32524461
- [Background] Lorimer PD, Motz BM, Kirks RC, Boselli DM, Walsh KK, Prabhu RS, Hill JS, Salo JC. Pathologic Complete Response Rates After Neoadjuvant Treatment in Rectal Cancer: An Analysis of the National Cancer Database. Ann Surg Oncol. 2017 Aug;24(8):2095-2103. doi: 10.1245/s10434-017-5873-8. Epub 2017 May 22. PMID 28534080
- [Background] Li Y, Wang J, Ma X, Tan L, Yan Y, Xue C, Hui B, Liu R, Ma H, Ren J. A Review of Neoadjuvant Chemoradiotherapy for Locally Advanced Rectal Cancer. Int J Biol Sci. 2016 Jul 17;12(8):1022-31. doi: 10.7150/ijbs.15438. eCollection 2016. PMID 27489505
- [Background] Bujko K, Wyrwicz L, Rutkowski A, Malinowska M, Pietrzak L, Krynski J, Michalski W, Oledzki J, Kusnierz J, Zajac L, Bednarczyk M, Szczepkowski M, Tarnowski W, Kosakowska E, Zwolinski J, Winiarek M, Wisniowska K, Partycki M, Beczkowska K, Polkowski W, Stylinski R, Wierzbicki R, Bury P, Jankiewicz M, Paprota K, Lewicka M, Cisel B, Skorzewska M, Mielko J, Bebenek M, Maciejczyk A, Kapturkiewicz B, Dybko A, Hajac L, Wojnar A, Lesniak T, Zygulska J, Jantner D, Chudyba E, Zegarski W, Las-Jankowska M, Jankowski M, Kolodziejski L, Radkowski A, Zelazowska-Omiotek U, Czeremszynska B, Kepka L, Kolb-Sielecki J, Toczko Z, Fedorowicz Z, Dziki A, Danek A, Nawrocki G, Sopylo R, Markiewicz W, Kedzierawski P, Wydmanski J; Polish Colorectal Study Group. Long-course oxaliplatin-based preoperative chemoradiation versus 5 x 5 Gy and consolidation chemotherapy for cT4 or fixed cT3 rectal cancer: results of a randomized phase III study. Ann Oncol. 2016 May;27(5):834-42. doi: 10.1093/annonc/mdw062. Epub 2016 Feb 15. PMID 26884592